CLINICAL TRIAL: NCT01306032
Title: Phase II Randomized Trial of ABT-888 in Combination With Metronomic Oral Cyclophosphamide in Refractory BRCA-Positive Ovarian, Primary Peritoneal, Ovarian High-Grade Serous Carcinoma, Fallopian Tube Cancer, or Triple-Negative Breast Cancer
Brief Title: Phase II ABT-888 With Cyclophosphamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 110080; 11-C-0080
Record Dates: First submitted 2011-02-26; First posted 2011-03-01 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Serous Carcinoma Cancer; Triple-Negative Breast Cancer; Fallopian Tube Cancer
Keywords: PARP Inhibitor; BRCA Mutations; DNA Damage Repair; Pharmacodynamics; Metronomic Cyclophosphamide; Ovarian Cancer; Breast Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms; Fallopian Tube Neoplasms; Breast Neoplasms | interventions — veliparib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide (Experimental): Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO) on a continuous schedule.
  Interventions: Drug: ABT-888; Drug: Cyclophosphamide
- Triple-negative Breast Cancer: Cyclophosphamide Alone (Experimental): Oral cyclophosphamide 50mg by mouth (PO) for 21 days. Participants in the cyclophosphamide alone arm crossed over to the ABT-888 plus cyclophosphamide arm at time of disease progression.
  Interventions: Drug: Cyclophosphamide
- BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide (Experimental): Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO) on a continuous schedule.
  Interventions: Drug: ABT-888; Drug: Cyclophosphamide
- BRCA- positive Ovarian Cancer: Cyclophosphamide Alone (Experimental): Oral cyclophosphamide 50mg by mouth (PO) for 21 days. Participants in the cyclophosphamide alone arm crossed over to the ABT-888 plus cyclophosphamide arm at time of disease progression.
  Interventions: Drug: Cyclophosphamide
- Non-Hodgkin's: ABT-888 + Cyclophosphamide (Experimental): Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO) on a continuous schedule.
  Interventions: Drug: ABT-888; Drug: Cyclophosphamide
- Non-Hodgkin's: Cyclophosphamide Alone (Experimental): Oral cyclophosphamide 50mg by mouth (PO) for 21 days. Participants in the cyclophosphamide alone arm crossed over to the ABT-888 plus cyclophosphamide arm at time of disease progression.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: ABT-888 — PARP enzymes are critical for maintaining genomic stability by regulating a variety of DNA repair mechanisms. Individuals with deleterious mutations in the BRCA1 or BRCA2 tumor suppressor genes have an increased risk of developing breast and ovarian cancers due to impaired or defective DNA damage repair; these individuals have an increased susceptibility to DNA-damaging agents and PARP inhibitors. Inhibition of PARP inhibits the repair of DNA damage caused by alkylating agents such as cyclophosphamide. Metronomic cyclophosphamide has demonstrated efficacy in several tumor types. The PARP inhibitor ABT-888 has been shown to potentiate the action of cyclophosphamide in xenograft models. This combination is well tolerated in a Phase I study and showing promising activity.
  Other Names: Veliparib
  Arms: BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide; Non-Hodgkin's: ABT-888 + Cyclophosphamide; Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide
Drug: Cyclophosphamide
  Other Names: Cytoxan

SUMMARY:
Background:

- The experimental cancer treatment drug ABT-888 (Veliparib) works by preventing deoxyribonucleic acid (DNA) repair in tumor cells. Cyclophosphamide is a cancer treatment drug that works by causing DNA damage in cells, including cancer cells, resulting in cell death. However, because cyclophosphamide has strong and unpleasant side effects, researchers are interested in finding drugs that can be given in combination with cyclophosphamide that will allow a lower dose of cyclophosphamide to be given with similar effects. The combination of ABT-88 and cyclophosphamide may be an effective treatment for some types of cancer, such as certain kinds of breast or ovarian cancer and non-Hodgkin's lymphoma that often do not respond to standard therapies.

Objectives:

- To evaluate the safety and effectiveness of ABT-888 and cyclophosphamide in ovarian and breast cancer and in non-Hodgkin's lymphoma that have not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with (1) (Breast cancer 1/2) BRCA1/2 ovarian cancer, primary peritoneal or ovarian high-grade carcinoma, or fallopian tube cancer; (2) triple-negative breast cancer (not responsive to hormone-related therapy); or (3) low grade non-Hodgkin's lymphoma.

Design:

* Participants will be screened with a full medical history and physical examination, blood and urine tests, and tumor imaging studies. Participants will be divided into two groups with different treatment subgroups.
* Group 1: Participants who have BRCA-positive ovarian cancer, primary peritoneal or ovarian high-grade serous carcinoma, or fallopian tube cancer
* Participants will receive either the combination of ABT-888 and cyclophosphamide, or cyclophosphamide alone.
* Participants will take the study drug by mouth once a day for 21-day cycles of treatment, and will keep a diary to record drug doses and any side effects.
* Participants will have clinic visits with blood and urine tests, imaging studies, and other examinations on days 1, 2, 7, and 14 of cycle 1, and on the first day of all other cycles.
* Group 2: Participants who have triple-negative breast cancer or non-Hodgkin's lymphoma
* Participants will receive either the combination of ABT-888 and cyclophosphamide, or cyclophosphamide alone.
* Participants will take the study drug by mouth once a day for 21-day cycles of treatment, and will keep a diary to record drug doses and any side effects.
* Participants will have clinic visits with blood and urine tests, imaging studies, and other examinations on days 1, 2, 7, and 14 of cycle 1, and on the first day of all other cycles.
* Participants receiving only cyclophosphamide who show signs of disease progression after tumor imaging studies can receive the combination of ABT-888 with cyclophosphamide.
* Treatment will continue as long as participants tolerate the drugs and the disease does not progress.

DETAILED DESCRIPTION:
Background:

* The poly (ADP-ribose) polymerase (PARP) family of enzymes is critical for maintaining genomic stability by regulating a variety of DNA repair mechanisms.
* Individuals with deleterious mutations in the BRCA1 or BRCA2 tumor suppressor genes have an increased risk of developing breast and ovarian cancers due to impaired or defective DNA damage repair; these individuals have an increased susceptibility to DNA-damaging agents and PARP inhibitors. Inhibition of PARP inhibits the repair of DNA damage caused by alkylating agents such as cyclophosphamide.
* Metronomic cyclophosphamide has demonstrated efficacy in several tumor types. The PARP inhibitor ABT-888 has been shown to potentiate the action of cyclophosphamide in xenograft models. This combination is well tolerated in a Phase I study and showing promising activity.

Objectives:

* Compare the response rate (complete response (CR) + partial response (PR)) of the combination of ABT-888 with metronomic oral cyclophosphamide to the response rate (CR+PR) of metronomic oral cyclophosphamide in patients with deleterious BRCA mutations and refractory ovarian cancer or patients with primary peritoneal or ovarian high-grade serous carcinoma or fallopian tube cancer.
* Compare the response rate (CR+PR) of the combination of ABT-888 with metronomic oral cyclophosphamide to the response rate (CR+PR) of single-agent oral cyclophosphamide in patients with triple-negative metastatic breast cancer, stratified for deleterious BRCA mutation.
* Compare the response rate (CR+PR) of the combination of ABT-888 with metronomic oral cyclophosphamide to the response rate (CR+PR) of single-agent metronomic oral cyclophosphamide in patients with refractory low-grade lymphomas.

Secondary Objectives:

- Determine PAR levels in tumor biopsies, evaluate in archival tissue whether patients tumors have mutations in genes involved in DNA damage repair (e.g., BRCA/Fanconi anemia/protein 53 (p53)), perform exploratory gene expression profiling to correlate PARP messenger ribonucleic acid (mRNA) levels or BRCA mutation status with response to therapy, count circulating tumor cells (CTCs), and determine H2AX levels in CTCs and tumor biopsies (National Cancer Institute (NCI) clinical center only).

Eligibility:

-Adults with refractory BRCA-positive ovarian cancer, primary peritoneal or ovarian high-grade serous carcinoma, fallopian tube cancer, triple-negative breast cancer, or low-grade lymphoid malignancies (non-Hodgkin's lymphoma) whose disease has progressed following at least one line of therapy.

Study Design:

* This is a randomized, multi-histology Phase II trial with patients enrolled into 3 cohorts: BRCA-positive ovarian cancer or primary peritoneal or ovarian high-grade serous carcinoma or fallopian tube cancer (A); triple-negative breast cancer (B); or low grade non-Hodgkin's lymphoma (C). Patients in cohort A will be randomized to the combination of ABT-888 with metronomic oral cyclophosphamide or metronomic oral cyclophosphamide alone. Patients in cohort B will be randomized to the combination of ABT-888 with metronomic oral cyclophosphamide or metronomic oral cyclophosphamide alone. Patients in cohort C will be randomized to the combination of ABT-888 with metronomic oral cyclophosphamide or metronomic oral cyclophosphamide alone.
* Cyclophosphamide (50 mg) and ABT-888 (60 mg) will be administered orally once a day, continuously in 21-day cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically documented:

  * BRCA-positive ovarian cancer (documented deleterious BRCA1/2 mutation or a BRCAPRO score of greater than or equal to 30%)
  * primary peritoneal or ovarian high-grade serous carcinoma or fallopian tube cancer (no requirement for BRCA status)
  * triple-negative breast cancer (documented estrogen receptor (ER) negative, progesterone receptor (PR) negative, and human epidermal growth factor receptor 2 (Her2/neu) negative from the original pathology report if considered adequate, or per The American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines (47, 48)) with metastasis to distant sites
  * Low-grade lymphoid malignancies (NHL), as described below, whose disease has progressed following at least one line of standard therapy:

    * Follicle center lymphoma, follicular or diffuse-recurrent/refractory
    * Marginal zone B-cell lymphoma: splenic, nodal, extranodal (this includes mucosa-associated lymphoid tissue (MALT)) - recurrent/refractory
    * Lymphoplasmacytic lymphoma - recurrent/refractory
    * Small lymphocytic lymphoma (SLL) (absolute lymphocytes count below 5,000)

Pathology must be confirmed by the registering institution. For patients who are eligible for the study due to a history of BRCA1/2 mutation, documented evidence of their mutation status must be provided prior to enrolling on the study.

* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* Any prior therapy or radiotherapy must have been completed greater than or equal to 4 weeks (greater than 6 weeks for nitrosoureas or mitomycin C) prior to enrollment on protocol, and the participant must have recovered to eligibility levels from prior toxicity. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study, and should have recovered to eligibility levels from any toxicities.
* Patients who have had prior treatment with any PARP inhibitors are eligible unless the PARP inhibitor was administered in combination with cyclophosphamide.
* Patients with bone metastases or hypercalcemia on bisphosphonate treatment are eligible to participate
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of ABT-888 in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I combination trials.
* Karnofsky performance status greater than or equal to 70%.
* Life expectancy greater than 3 months.
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/microL (mcL)
  * platelets greater than or equal to 100,000/microL (mcL)
  * total bilirubin less than 1.5 times institutional upper limit of normal
  * Aspartate aminotransaminase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransaminase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * creatinine less than 1.5 times institutional upper limit of normal

OR

--creatinine clearance greater than or equal to 60 mL/min for patients with creatinine

levels greater than or equal to 1.5 times institutional upper limit of normal.

* The effects of ABT-888 on the developing human fetus are unknown. For this reason and because cyclophosphamide hydrochloride is known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (abstinence; female use of hormonal methods, or barrier methods of birth control; male use of a condom) prior to study entry, for the duration of study participation, and for 3 months after completion of study. Because there is a risk for adverse events in nursing infants secondary to treatment of the mother with cyclophosphamide, breastfeeding should be discontinued while the patient is on this trial and for 30 days after completion of treatment on this trial. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Women who are pregnant or breastfeeding.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with germ cell and borderline ovarian epithelial tumors.
* Patients who have received prior cyclophosphamide should not be excluded solely because of receiving prior cyclophosphamide.
* Patients with history of central nervous system (CNS) metastases who have received treatment and who have been on stable doses of anti-seizure medicine and had no seizures x 3 months will be eligible.
* Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, and active peptic ulcer disease) are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded, as are any patients who cannot swallow the capsule whole. Capsules must not be crushed or chewed; nasogastric or gastrostomy tube (G-tube) administration is not allowed.

INCLUSION OF WOMEN AND MINORITIES:

-Men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-01-12 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (10):
- United States (9):
  - University of California, Davis, Davis, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data are being shared with this CT.gov report and two peer-reviewed publications. There is no plan to share individual patient results.

REFERENCES:
- [Background] Donawho CK, Luo Y, Luo Y, Penning TD, Bauch JL, Bouska JJ, Bontcheva-Diaz VD, Cox BF, DeWeese TL, Dillehay LE, Ferguson DC, Ghoreishi-Haack NS, Grimm DR, Guan R, Han EK, Holley-Shanks RR, Hristov B, Idler KB, Jarvis K, Johnson EF, Kleinberg LR, Klinghofer V, Lasko LM, Liu X, Marsh KC, McGonigal TP, Meulbroek JA, Olson AM, Palma JP, Rodriguez LE, Shi Y, Stavropoulos JA, Tsurutani AC, Zhu GD, Rosenberg SH, Giranda VL, Frost DJ. ABT-888, an orally active poly(ADP-ribose) polymerase inhibitor that potentiates DNA-damaging agents in preclinical tumor models. Clin Cancer Res. 2007 May 1;13(9):2728-37. doi: 10.1158/1078-0432.CCR-06-3039. PMID 17473206
- [Background] Shiobara M, Miyazaki M, Ito H, Togawa A, Nakajima N, Nomura F, Morinaga N, Noda M. Enhanced polyadenosine diphosphate-ribosylation in cirrhotic liver and carcinoma tissues in patients with hepatocellular carcinoma. J Gastroenterol Hepatol. 2001 Mar;16(3):338-44. doi: 10.1046/j.1440-1746.2001.02378.x. PMID 11339428
- [Background] Tomoda T, Kurashige T, Moriki T, Yamamoto H, Fujimoto S, Taniguchi T. Enhanced expression of poly(ADP-ribose) synthetase gene in malignant lymphoma. Am J Hematol. 1991 Aug;37(4):223-7. doi: 10.1002/ajh.2830370402. PMID 1907096
- [Result] Kummar S, Oza AM, Fleming GF, Sullivan DM, Gandara DR, Naughton MJ, Villalona-Calero MA, Morgan RJ Jr, Szabo PM, Youn A, Chen AP, Ji J, Allen DE, Lih CJ, Mehaffey MG, Walsh WD, McGregor PM 3rd, Steinberg SM, Williams PM, Kinders RJ, Conley BA, Simon RM, Doroshow JH. Randomized Trial of Oral Cyclophosphamide and Veliparib in High-Grade Serous Ovarian, Primary Peritoneal, or Fallopian Tube Cancers, or BRCA-Mutant Ovarian Cancer. Clin Cancer Res. 2015 Apr 1;21(7):1574-82. doi: 10.1158/1078-0432.CCR-14-2565. Epub 2015 Jan 14. PMID 25589624
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0080.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Triple-negative breast cancer participants were enrolled but three did not start the study (two withdrew, 1 progressed).
Groups:
- BRCA-positive Ovarian Cancer: Cyclophosphamide Alone; Non-Hodgkin's: Cyclophosphamide Alone: Oral cyclophosphamide 50mg by mouth (PO) for 21 days. Participants in the cyclophosphamide alone arm crossed over to the ABT-888 plus cyclophosphamide arm at time of disease progression.
Period: First Intervention
Arm/Group | Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide | Triple-negative Breast Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | Non-Hodgkin's: ABT-888 + Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
Started | 22 | 20 (Not all participants on the Cyclophosphamide Alone Arm met eligibility criteria to crossover.) | 37 | 38 (Not all participants on the Cyclophosphamide Alone Arm met eligibility criteria to crossover.) | 2 | 2
Completed | 21 | 18 | 35 | 37 | 0 | 0
Not Completed | 1 | 2 | 2 | 1 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Ineligible | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 2 | 0
Period: Disease Progression/Crossover
Arm/Group | Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide | Triple-negative Breast Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | Non-Hodgkin's: ABT-888 + Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
Started | 0 | 16 | 0 | 29 | 0 | 0
Completed | 0 | 14 | 0 | 26 | 0 | 0
Not Completed | 0 | 2 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — other/symptomatic progression | 0 | 2 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide; BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide; Non-Hodgkin's: ABT-888 + Cyclophosphamide: Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO).
- Triple-negative Breast Cancer: Cyclophosphamide Alone; BRCA-positive Ovarian Cancer: Cyclophosphamide Alone; Non-Hodgkin's: Cyclophosphamide Alone: Oral cyclophosphamide 50mg by mouth (PO) for 21 days.
- Total: Total of all reporting groups
Arm/Group | Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide | Triple-negative Breast Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | Non-Hodgkin's: ABT-888 + Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone | Total
Number analyzed (Participants) | 25 | 20 | 37 | 38 | 2 | 2 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 28 | 29 | 1 | 2 | 96
  >=65 years | 5 | 4 | 9 | 9 | 1 | 0 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10) | 53 (13) | 57 (10) | 58 (10) | 70 (24) | 56 (6) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 37 | 38 | 1 | 2 | 123
  Male | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 22 | 17 | 36 | 35 | 1 | 2 | 113
  Unknown or Not Reported | 2 | 1 | 0 | 2 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 1 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 0 | 0 | 0 | 0 | 10
  White | 16 | 15 | 35 | 37 | 2 | 2 | 107
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 17 | 23 | 23 | 2 | 2 | 89
  Canada | 3 | 3 | 14 | 15 | 0 | 0 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Overall Response Rate
Description: Complete response (CR) + partial response (PR)) of the combination of ABT-888 with metronomic oral cyclophosphamide to the response rate (CR+PR) of metronomic oral cyclophosphamide in patients with deleterious BRCA mutations and refractory ovarian cancer or patients with primary peritoneal or ovarian high-grade serous carcinoma or fallopian tube cancer. CR + PR was determined by the Response Evaluation Criteria in Solid Tumors (RECIST). CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm). Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: an average of 126 days for ovarian; 71 days for TNBC; for crossover intervention, pts stayed on study for an avg of 134 days for ovarian; 50 days for TNBC.
Population: Participants evaluable for response.
Measure: Number; unit: percentage of participants
Groups:
- Triple-negative Breast Cancer: Crossover; BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide; BRCA-positive Ovarian Cancer: Crossover: Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO) on a continuous schedule.
Arm/Group | Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide | Triple-negative Breast Cancer: Cyclophosphamide Alone | Triple-negative Breast Cancer: Crossover | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: Crossover
Number analyzed (Participants) | 21 | 18 | 16 | 34 | 36 | 29
percentage of participants | 9.5 | 5.6 | 0 | 11.8 | 19.4 | 3.4

2. Primary Outcome: Progression Free Survival
Description: Time to progression for each participant for the initial intervention.
Time Frame: Ovarian cancer patients stayed on study for an average of 126 days and triple-negative breast cancer patients for an average of 71 days.
Population: Participants evaluable for response.
Measure: Median (Full Range); unit: Cycles of therapy
Arm/Group | Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide | Triple-negative Breast Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone
Number analyzed (Participants) | 21 | 18 | 34 | 36
Cycles of therapy | 3 [1 to 3] | 2 [1 to 9] | 3 [1 to 39] | 3 [1 to 32]
Statistical Analysis 1: Comparison: Triple-negative Breast Cancer: ABT-888 + Cyclophosphamide vs Triple-negative Breast Cancer: Cyclophosphamide Alone; Test type: Superiority or Other; p = 0.034, Log Rank
Statistical Analysis 2: Comparison: BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide vs BRCA-positive Ovarian Cancer: Cyclophosphamide Alone; Test type: Superiority or Other; p = 0.68, Log Rank

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: up to 30 days following the last dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- BRCA-positive Ovarian Cancer: ABT-888 & Cyclophosphamide; BRCA-positive Ovarian Cancer: Crossover; Triple-negative Breast Cancer: Crossover; Non-Hodgkin's: ABT-888 & Cyclophosphamide: Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO) on a continuous schedule.
- Triple-negative Breast Cancer: Cyclophosphamide & ABT-888: Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth on a continuous schedule.
Arm/Group | BRCA-positive Ovarian Cancer: ABT-888 & Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: Crossover | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 | Triple-negative Breast Cancer: Cyclophosphamide Alone | Triple-negative Breast Cancer: Crossover | Non-Hodgkin's: ABT-888 & Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
Number analyzed (Participants) | 37 | 38 | 29 | 21 | 18 | 16 | 2 | 1
Participants | 28 | 24 | 29 | 14 | 4 | 6 | 0 | 1

4. Secondary Outcome: Change in Poly-ADP Ribose (PAR) Concentration Levels From Baseline
Description: PAR levels (in pg/μg protein) were assessed in peripheral blood mononuclear cells (PBMCs) by immunoassay to assess poly (ADP-ribose) polymerase (PARP) activity. Significant inhibition of PARP activity is associated with 50% or greater reduction in PAR levels.
Time Frame: At baseline (t=0h) and 4h post drug administration (t=4h)
Population: Patients with PBMCs data pre- and post-drug administration, and with PAR levels above the lower limit of quantitation (LLOQ) of 23 pg/μg protein were analyzed.
Measure: Mean (Full Range); unit: pg/μg protein
Arm/Group | BRCA-positive Ovarian Cancer: ABT-888 & Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: Crossover | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 | Triple-negative Breast Cancer: Cyclophosphamide Alone | Triple-negative Breast Cancer: Crossover | Non-Hodgkin's: ABT-888 & Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
Number analyzed (Participants) | 10 | 0 | 11 | 4 | 0 | 2 | 0 | 0
pg/μg protein | -81 [-93 to -48] |  | -88 [-97 to -68] | -74 [-83 to -65] |  | -85 [-85 to -85] |  |

5. Secondary Outcome: Change in ϓH2AX- Positive Circulating Tumor Cells (CTCs) in Whole Blood
Description: Number of CTCs (evaluable defined as ≥ 6 CTCs) were measured in whole blood during the course of treatment to determine drug-induced deoxyribonucleic acid damage in tumor cells.
Time Frame: At baseline (t=0h) and 24h post drug administration (t=24h)
Population: Patients with sufficient CTC counts (defined as ≥6 total CTCs) pre- and post-drug administration were analyzed.
Measure: Mean (Full Range); unit: ϓH2AX- Positive CTCs
Arm/Group | BRCA-positive Ovarian Cancer: ABT-888 & Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: Crossover | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 | Triple-negative Breast Cancer: Cyclophosphamide Alone | Triple-negative Breast Cancer: Crossover | Non-Hodgkin's: ABT-888 & Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
ϓH2AX- Positive CTCs |  |  | 400 [400 to 400] | 200 [200 to 200] |  | 9.5 [-38 to 57] |  |

6. Secondary Outcome: Number of Participants With Deleterious Mutations in DNA Repair Genes
Description: Gene expression profiling was performed in archival tumor tissue for a panel of 211 genes using deoxyribonucleic acid (DNA) array to determine deleterious mutations (i.e. nonsynonymous mutations at coding regions) of genes. Sequences were mapped to human genome reference hg19. Variants were identified with VarScan, annotated with AVIA, and masked to the exonic or exonic:splicing regions of the 211 interrogated DNA repair genes, with nonsynonymous/frameshift/stop-gain/stop-loss variants that have a population frequency of 1% or less in either 1000G (2014_04) or the ExomeSequencingProject (ESP6500si_all) with a minimum variant frequency of 10% and at least 20 reads. Lastly, variants were manually inspected for known platform and mapping errors.
Time Frame: Optional tumor biopsies were performed prior to start of treatment (baseline) and 6 months
Population: Patients with sufficient tumor content in archival tissue (defined as ≥70% tumor after macrodissection) were analyzed for genetic alterations in DNA repair genes by whole-exome sequencing.
Measure: Count of Participants; unit: Participants
Arm/Group | BRCA-positive Ovarian Cancer: ABT-888 & Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: Crossover | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 | Triple-negative Breast Cancer: Cyclophosphamide Alone | Triple-negative Breast Cancer: Crossover | Non-Hodgkin's: ABT-888 & Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
Number analyzed (Participants) | 28 | 0 | 27 | 0 | 0 | 0 | 0 | 0
Participants | 28 |  | 27 |  |  |  |  |

ADVERSE EVENTS:
Time Frame: up to 30 days following the last dose of study drug.
Description: Adverse events were categorized by treatment (initial vs. crossover treatment arms) rather than indication as this was how we analyzed the data.
Groups:
- Triple-negative Breast Cancer: Cyclophosphamide & ABT-888; Triple-negative Breast Cancer: Crossover; Non-Hodgkin's: ABT-888 + Cyclophosphamide: Oral cyclophosphamide 50mg by mouth (PO) for 21 days and oral ABT-888 60mg by mouth (PO) on a continuous schedule.
Arm/Group | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone | BRCA-positive Ovarian Cancer: Crossover | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 | Triple-negative Breast Cancer: Cyclophosphamide Alone | Triple-negative Breast Cancer: Crossover | Non-Hodgkin's: ABT-888 + Cyclophosphamide | Non-Hodgkin's: Cyclophosphamide Alone
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/38 | 0/29 | 0/21 | 0/18 | 0/16 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/37 | 0/38 | 0/29 | 2/21 | 0/18 | 1/16 | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 28/37 | 24/38 | 29/29 | 14/21 | 4/18 | 6/16 | 0/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide (N=37) | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone (N=38) | BRCA-positive Ovarian Cancer: Crossover (N=29) | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 (N=21) | Triple-negative Breast Cancer: Cyclophosphamide Alone (N=18) | Triple-negative Breast Cancer: Crossover (N=16) | Non-Hodgkin's: ABT-888 + Cyclophosphamide (N=2) | Non-Hodgkin's: Cyclophosphamide Alone (N=1)
Lymphopenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Death Not Associated with CTCAE: Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRCA-positive Ovarian Cancer: ABT-888 + Cyclophosphamide (N=37) | BRCA-positive Ovarian Cancer: Cyclophosphamide Alone (N=38) | BRCA-positive Ovarian Cancer: Crossover (N=29) | Triple-negative Breast Cancer: Cyclophosphamide & ABT-888 (N=21) | Triple-negative Breast Cancer: Cyclophosphamide Alone (N=18) | Triple-negative Breast Cancer: Crossover (N=16) | Non-Hodgkin's: ABT-888 + Cyclophosphamide (N=2) | Non-Hodgkin's: Cyclophosphamide Alone (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 | 0 | 0 | 1 (2) | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0
Oral mucositis (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 9 (16) | 2 (6) | 9 (9) | 3 (3) | 3 (5) | 2 (4) | 0 | 0
Leucopenia (Investigations) | 12 (27) | 6 (14) | 8 (9) | 4 (8) | 0 | 0 | 0 | 0
Neutropenia (Investigations) | 7 (22) | 1 (2) | 4 (4) | 1 (6) | 0 | 0 | 0 | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 2 (2) | 0 | 0 | 0 | 0
Pelvic infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 (4) | 3 (3) | 5 (5) | 0 | 2 (2) | 3 (3) | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Hyperchloremia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
ALT increased (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Lymphopenia (Investigations) | 23 (62) | 16 (33) | 18 (36) | 9 (21) | 3 (3) | 3 (4) | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Psychiatric disorders, other (tearfulness) (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
AST increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0
PTT prolonged (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0
ALP increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Thrombocytopenia (Investigations) | 3 (5) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No